CLINICAL TRIAL: NCT03694561
Title: Developing a Management Approach for Patients With "Late-Onset" Pompe Disease GAA Variant Identified by Newborn Screening
Brief Title: Developing a Management Approach for Patients With "Late-Onset" Pompe Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00100223
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Pompe Disease; Pompe Disease (Late-onset); GAA Deficiency
Keywords: Pompe disease; Glycogen Storage Disease Type II; Acid Maltase Deficiency; Acid Alpha-Glucosidase Deficiency; Alglucosidase alfa; Newborn Screening
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Late-Onset Pompe disease: Individuals with a confirmed diagnosis of Late-Onset Pompe disease via NBS
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — This study is a systematic investigation of the natural history of late-onset Pompe disease in infancy and childhood

SUMMARY:
This is an observational study with no study related treatment of interventions. The purpose of the study is to investigate and document disease specific clinical symptoms in newborns, infants and children with Pompe disease without cardiomyopathy identified in newborn screening(NBS).

There will be baseline, months 6 and months 12 visits for infants and newborns (infants study). For children of ages 24 months to 54 months, there will be baseline, year 1 and year 2 visits (children study).

The study has four goals:

1. To study and record disease specific clinical symptoms in newborns, infants and children with Pompe disease without cardiomyopathy (disease of the heart muscle) in the first year of life identified through newborn screening (NBS)
2. To devise an approach to characterize early musculoskeletal (muscles and joints) involvement in subjects with the "late-onset" GAA variant identified by NBS including ability to collect research information via virtual health platforms.
3. To determine criteria to start preventative therapies including enzyme replacement therapy (ERT) in patients with clinical features of Pompe disease identified via NBS
4. To document parental coping and anxiety/emotional distress overtime using quality of life questionnaires after a child is diagnosed with late onset Pompe disease via NBS

DETAILED DESCRIPTION:
Late-Onset Pompe Disease(LOPD) is an inherited disorder caused by lack of or defect in the enzyme acid alpha-glucosidase (GAA). GAA enzyme deficiency causes glycogen to build up and damage cells throughout the body, especially in the heart and muscles. In LOPD, subtle and overt disease-specific features may go unrecognized in childhood without vigilant clinical examination and assessments with appropriate functional tests. In our clinical experience, children with the "late-onset" GAA variant may present much earlier in life and adult patients with LOPD consistently report a much earlier symptom onset and a significant diagnostic delay. These patients have shown improvement after initiation of ERT but have motor impairments adversely affecting their quality of life and growth from early childhood. Therefore, earlier diagnosis and initiation of ERT is crucial in these patients. Instituting ERT at an ideal time may prevent/reduce these irreversible musculoskeletal impairments and lead to a better quality of life and less disease burden as these children age.

Our team of Pompe disease experts will perform detailed clinical evaluations, physical therapy evaluations, cardiac assessments, speech and swallow evaluations, biochemical tests, sleep questionnaire, and hearing assessments on these patients. These assessments will allow use to capture and describe the earlier clinical phenotype in these patients and provide insights into the early signs and symptoms of LOPD.This study will provide and evidence-based approach to clinical management of newborns with LOPD to primary care physicians and geneticists, leading to improves patient outcomes.

The investigators will enroll 20 infants and children at Duke that has screened for LOPD. This study involves minimal risk to the patient and offers a potential benefit of improved disease management. For infants, the initial visit will be as soon as possible after a confirmed LOPD diagnosis and follow up visits will be at 6 months and 12 months. The investigators will continue to gather clinical information on patients and monitor clinical status beyond assessment at three time points. For children of ages 24 months to 54 months, there will be baseline, year 1 and year 2 visits.

The study has four goals:

1. To study and record disease specific clinical symptoms in newborns, infants and children with Pompe disease without cardiomyopathy (disease of the heart muscle) in the first year of life identified through newborn screening (NBS)
2. To devise an approach to characterize early musculoskeletal (muscles and joints) involvement in subjects with the "late-onset" GAA variant identified by NBS including ability to collect research information via virtual health platforms.
3. To determine criteria to start preventative therapies including enzyme replacement therapy (ERT) in patients with clinical features of Pompe disease identified via NBS
4. To document parental coping and anxiety/emotional distress overtime using quality of life questionnaires after a child is diagnosed with late onset Pompe disease via NBS

ELIGIBILITY:
Inclusion Criteria:

* Subject has been diagnosed via newborn screening
* Subject has a confirmed and documented diagnosis of Pompe disease and absence of cardiac involvement
* Subject has predicted "late-onset" GAA variants such as c.-32-13T>G, c.2188G>T, c.1935C>A, c.1726G>A, c.118C>T etc. in homozygosity or compound heterozygosity
* Subject must be between 3 and 20 months for infant study or between 24 and 54 months (+/- 3 months) for children study at time of enrollment.

Ages: 3 Months to 54 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants who have been diagnosed with Late-Onset Pompe Disease via Newborn Screening (NBS)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Medical records will be tracked for up to 4.5 years to document subtle musculoskeletal signs of Pompe disease. | 4.5 years
  This outcome measure will be tested individually by a formal physical therapy assessment, Alberta Infant Motor Scale (AIMS), Gross Motor Functional Measure (GMFM), Hammersmith Functional Motor Scale Expanded(HFMSE),Modified Hammersmith Functional Motor Scale Extend(MHMFS-EXTEND), and Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders(CHOP INTEND) to give a combined assessment score.
Medical records will be tracked for up to 4.5 years years to document Pompe-specific clinical symptoms. | 4.5 years
  This outcome measure will be tested individually by physical examination, nutritional evaluation and functional assessment to give a combined analysis of Pompe-specific symptoms.
Medical records will be tracked for 4.5 years to document elevation in Pompe-specific biomarkers from blood and urine samples. | 4.5 years
  This outcome measure will be tested by comparing lab results to lab-specific ranges.

SECONDARY OUTCOMES:
Medical records will be tracked for 4.5 years to document sleep quality. | 4.5 years
  This outcome measure will be tested qualitatively by questionnaire.
Medical records will be tracked for 4.5 years to document auditory capacity. | 4.5 years
  This outcome measure will be tested individually by visual reinforcement audiology (VRA) and distortion product optoacoustic emissions (DPOAE) to give a combined assessment score.
Medical records will be tracked for 4.5 years to document cardiac involvement. | 4.5 years
  This outcome measure will be analyzed by echocardiogram and electrocardiogram results.
Medical records will be tracked for 4.5 years to document muscle architecture of the calves, para-spinal muscles and tongue | 4.5 years
  This outcome measure will be tested qualitatively by simple ultrasound examination.
Medical records will be tracked for 4.5 years to document speech and swallow progression | 4.5 years
  This outcome measure will be tested individually by using videofluoroscopic study, Preschool Language Scale-Fourth Edition(PLS4), Receptive-Expressive Emergent Language Test Third Edition(REEL3), Pediatric Eating Assessment Tool (PEDI EAT-10), Functional Oral Intake Scale(FOIS) and serial photographs to give a combined assessment score.
Change in parental coping overtime using quality of life questionnaires after a child is diagnosed with late onset Pompe disease via NBS. | yearly, up to 4.5 years
  BRIEF COPE is completed by the patient's parent or guardian. BRIEF COPE is rated on a scale of 1-4 with 1 = 'I haven't been doing this at all' and 4 = 'I've been doing this a lot'.
Change in parent's emotional distress overtime using PROMIS questionnaire | yearly, up to 4.5 years
  The PROMIS questionnaire is completed by the patient's parent or guardian. Emotional distress is rated on a scale of 1-5 with 1=never and 5=always.

CONTACTS AND LOCATIONS:
Overall Officials: Priya Kishnani, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chien YH, Hwu WL, Lee NC. Pompe disease: early diagnosis and early treatment make a difference. Pediatr Neonatol. 2013 Aug;54(4):219-27. doi: 10.1016/j.pedneo.2013.03.009. Epub 2013 Apr 28. PMID 23632029
- [Background] Chien YH, Lee NC, Thurberg BL, Chiang SC, Zhang XK, Keutzer J, Huang AC, Wu MH, Huang PH, Tsai FJ, Chen YT, Hwu WL. Pompe disease in infants: improving the prognosis by newborn screening and early treatment. Pediatrics. 2009 Dec;124(6):e1116-25. doi: 10.1542/peds.2008-3667. PMID 19948615
- [Background] Chien YH, Chiang SC, Zhang XK, Keutzer J, Lee NC, Huang AC, Chen CA, Wu MH, Huang PH, Tsai FJ, Chen YT, Hwu WL. Early detection of Pompe disease by newborn screening is feasible: results from the Taiwan screening program. Pediatrics. 2008 Jul;122(1):e39-45. doi: 10.1542/peds.2007-2222. Epub 2008 Jun 2. PMID 18519449
- [Background] Chien YH, Lee NC, Chen CA, Tsai FJ, Tsai WH, Shieh JY, Huang HJ, Hsu WC, Tsai TH, Hwu WL. Long-term prognosis of patients with infantile-onset Pompe disease diagnosed by newborn screening and treated since birth. J Pediatr. 2015 Apr;166(4):985-91.e1-2. doi: 10.1016/j.jpeds.2014.10.068. Epub 2014 Nov 4. PMID 25466677
- [Background] Feeney EJ, Austin S, Chien YH, Mandel H, Schoser B, Prater S, Hwu WL, Ralston E, Kishnani PS, Raben N. The value of muscle biopsies in Pompe disease: identifying lipofuscin inclusions in juvenile- and adult-onset patients. Acta Neuropathol Commun. 2014 Jan 2;2:2. doi: 10.1186/2051-5960-2-2. PMID 24383498
- [Background] Hagemans ML, Hop WJ, Van Doorn PA, Reuser AJ, Van der Ploeg AT. Course of disability and respiratory function in untreated late-onset Pompe disease. Neurology. 2006 Feb 28;66(4):581-3. doi: 10.1212/01.wnl.0000198776.53007.2c. PMID 16505317
- [Background] Hagemans ML, Winkel LP, Van Doorn PA, Hop WJ, Loonen MC, Reuser AJ, Van der Ploeg AT. Clinical manifestation and natural course of late-onset Pompe's disease in 54 Dutch patients. Brain. 2005 Mar;128(Pt 3):671-7. doi: 10.1093/brain/awh384. Epub 2005 Jan 19. PMID 15659425
- [Background] Kishnani PS, Hwu WL, Mandel H, Nicolino M, Yong F, Corzo D; Infantile-Onset Pompe Disease Natural History Study Group. A retrospective, multinational, multicenter study on the natural history of infantile-onset Pompe disease. J Pediatr. 2006 May;148(5):671-676. doi: 10.1016/j.jpeds.2005.11.033. PMID 16737883
- [Background] Kishnani PS, Steiner RD, Bali D, Berger K, Byrne BJ, Case LE, Crowley JF, Downs S, Howell RR, Kravitz RM, Mackey J, Marsden D, Martins AM, Millington DS, Nicolino M, O'Grady G, Patterson MC, Rapoport DM, Slonim A, Spencer CT, Tifft CJ, Watson MS. Pompe disease diagnosis and management guideline. Genet Med. 2006 May;8(5):267-88. doi: 10.1097/01.gim.0000218152.87434.f3. No abstract available. PMID 16702877
- [Background] Kroos MA, Pomponio RJ, Hagemans ML, Keulemans JL, Phipps M, DeRiso M, Palmer RE, Ausems MG, Van der Beek NA, Van Diggelen OP, Halley DJ, Van der Ploeg AT, Reuser AJ. Broad spectrum of Pompe disease in patients with the same c.-32-13T->G haplotype. Neurology. 2007 Jan 9;68(2):110-5. doi: 10.1212/01.wnl.0000252798.25690.76. PMID 17210890
- [Background] Laforet P, Laloui K, Granger B, Hamroun D, Taouagh N, Hogrel JY, Orlikowski D, Bouhour F, Lacour A, Salort-Campana E, Penisson-Besnier I, Sacconi S, Zagnoli F, Chapon F, Eymard B, Desnuelle C, Pouget J; French Pompe Registry Study Group. The French Pompe registry. Baseline characteristics of a cohort of 126 patients with adult Pompe disease. Rev Neurol (Paris). 2013 Aug-Sep;169(8-9):595-602. doi: 10.1016/j.neurol.2013.07.002. Epub 2013 Sep 3. PMID 24008051
- [Background] Rairikar MV, Case LE, Bailey LA, Kazi ZB, Desai AK, Berrier KL, Coats J, Gandy R, Quinones R, Kishnani PS. Insight into the phenotype of infants with Pompe disease identified by newborn screening with the common c.-32-13T>G "late-onset" GAA variant. Mol Genet Metab. 2017 Nov;122(3):99-107. doi: 10.1016/j.ymgme.2017.09.008. Epub 2017 Sep 19. PMID 28951071
- [Background] Wokke JH, Escolar DM, Pestronk A, Jaffe KM, Carter GT, van den Berg LH, Florence JM, Mayhew J, Skrinar A, Corzo D, Laforet P. Clinical features of late-onset Pompe disease: a prospective cohort study. Muscle Nerve. 2008 Oct;38(4):1236-45. doi: 10.1002/mus.21025. PMID 18816591